CLINICAL TRIAL: NCT01657396
Title: Implementation and Evaluation of Revised Protocols for Oral Hygiene for Mechanically Ventilated Patients in Alberta Health Services Calgary Region - a Pilot Project.
Brief Title: Implementation and Evaluation of Revised Protocols for Oral Hygiene for Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Sage Products, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Dan Zuege, Clinical Associate Professor of Medicine, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23068
Record Dates: First submitted 2012-07-25; First posted 2012-08-06 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Ventilator Associated Pneumonia; Oral Hygiene
Keywords: Oral Care; Oral Hygiene; Intensive Care; Mechanical Ventilation; Chlorhexidine
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Oral Hygiene (Active Comparator): Oral hygiene provided by current local standard of care - minimum q2h mouthcare with a green Toothette swab dipped in sterile water, with excess liquid aspirated using a Yankauer suction. Brushing of teeth (if applicable) with a toothbrush and standard toothpaste q12h. Replacement of Yankauer suction device daily.
  Interventions: Procedure: Standard Oral Hygiene
- SAGE Q-care q2 (Active Comparator): Oral hygiene provided with a commercial pre-packaged product (SAGE Q-care q2 Oral Cleansing and Suctioning System) - minimum q2h mouthcare using the supplied applicator swabs and covered Yankauer suction device using supplied Perox-A-Mint (a hydrogen peroxide based oral hygiene solution) alternating with alcohol-free mouthwash. Brushing of teeth (if applicable) with supplied applicator using Antiplaque solution (a cetylpyridinium based solution) q12h. Use of a new kit (which includes new covered Yankauer suction device) daily.
  Interventions: Procedure: SAGE Q-care q2
- SAGE Q-care q2 with Chlorhexidine (Active Comparator): Oral hygiene provided with a commercial pre-packaged product with chlorhexidine (SAGE Q-care Rx q2 Oral Cleansing and Suctioning System with CHG) - minimum q2h mouthcare using the supplied applicator swabs and covered Yankauer suction device using supplied Perox-A-Mint (a hydrogen peroxide based oral hygiene solution) alternating with alcohol-free mouthwash. Brushing of teeth (if applicable) with supplied applicator using chlorhexidine oral rinse (solution containing 0.12% chlorhexidine) q12h. Use of a new kit (which includes new covered Yankauer suction device) daily.
  Interventions: Procedure: SAGE Q-care q2 with Chlorhexidine

INTERVENTIONS:
Procedure: Standard Oral Hygiene — Current local standard of care - minimum q2h mouthcare with a green Toothette swab dipped in sterile water, with excess liquid aspirated using a Yankauer suction. Brushing of teeth (if applicable) with a toothbrush and standard toothpaste q12h. Replacement of Yankauer suction device daily.
  Arms: Standard Oral Hygiene
Procedure: SAGE Q-care q2 — Oral hygiene provided with a commercial pre-packaged product (SAGE Q-care q2 Oral Cleansing and Suctioning System) - minimum q2h mouthcare using the supplied applicator swabs and covered Yankauer suction device using supplied Perox-A-Mint (a hydrogen peroxide based oral hygiene solution) alternating with alcohol-free mouthwash. Brushing of teeth (if applicable) with supplied applicator using Antiplaque solution (a cetylpyridinium based solution) q12h. Use of a new kit (which includes new covered Yankauer suction device) daily.
  Arms: SAGE Q-care q2
Procedure: SAGE Q-care q2 with Chlorhexidine — Oral hygiene provided with a commercial pre-packaged product with chlorhexidine (SAGE Q-care Rx q2 Oral Cleansing and Suctioning System with CHG) - minimum q2h mouthcare using the supplied applicator swabs and covered Yankauer suction device using supplied Perox-A-Mint (a hydrogen peroxide based oral hygiene solution) alternating with alcohol-free mouthwash. Brushing of teeth (if applicable) with supplied applicator using chlorhexidine oral rinse (solution containing 0.12% chlorhexidine) q12h. Use of a new kit (which includes new covered Yankauer suction device) daily.
  Arms: SAGE Q-care q2 with Chlorhexidine

SUMMARY:
The primary objective of this study is to evaluate the effectiveness and feasibility of the implementation of revised standards of care for oral hygiene (SAGE Q-care q2 Oral Cleansing and Suctioning System with and without chlorhexidine gluconate) relative to the current routine standard of care in mechanically ventilated patients admitted to the adult Intensive Care Units in Alberta Health Services Calgary Zone. This pilot study will evaluate the feasibility of performing a larger definitive study. The primary assessment of effectiveness for the definitive study will be the proportion of patients who develop ventilator-associated pneumonia.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effectiveness and feasibility of the implementation of revised standards of care for oral hygiene (SAGE Q-care q2 Oral Cleansing and Suctioning System with and without chlorhexidine gluconate) relative to the current routine standard of care in mechanically ventilated patients admitted to the adult Intensive Care Units in Alberta Health Services Calgary Zone. This pilot study will evaluate the feasibility of performing a larger definitive study. The primary assessment of effectiveness for the definitive study will be the proportion of patients who develop ventilator-associated pneumonia.

150 subjects will be randomly assigned using sealed opaque envelopes to one of three groups (Oral hygiene provided via the current local standard of care; Oral hygiene provided with a commercial packaged product (SAGE Q-care q2 Oral Cleansing and Suctioning System); Oral hygiene provided with a similar commercial packaged product with added chlorhexidine rinses twice daily (SAGE 24-Hour Suction Systems with chlorhexidine gluconate). Subjects will be provided the assigned method of oral hygiene by the bedside nurses from the time of ICU admission to the time of ICU discharge.

Key measurements include the acquisition of ventilator-associated pneumonia; the documented frequency of provision of oral care; the state of oral hygiene evaluated by recorded oral hygiene scores; duration of mechanical ventilation; ICU and hospital lengths of stay; ICU and hospital survival; Antimicrobial utilization; and the acquisition of antimicrobial resistant microbes.

For comparison of outcomes, means (with standard deviations) and medians (with interquartile ranges) will be reported for normally distributed and skewed variables respectively, and will be compared among the three groups using ANOVA or Kruskal-Wallis tests, respectively. Only the first episode of VAP in a patient will be evaluated. Given the small size of this pilot study, no interim or subgroup analyses are planned.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years old)
* Newly admitted to the intensive care unit
* Receiving invasive mechanical ventilation via a endotracheal tube or tracheostomy

Exclusion Criteria:

* Under the age of 18
* Documented allergy to chlorhexidine
* Contraindication to the provision of standard oral hygiene (eg. recent oropharyngeal surgery or a defined surgical limitation to oral care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Ventilator-associated pneumonia | Subjects will be assessed for this outcome from the date of randomization until discharge from the ICU (up to 30 days post-randomization)

SECONDARY OUTCOMES:
Frequency of documented oral care procedures | The frequency of oral care procedures will be assessed daily from the date of randomization until discharge from the ICU (up to 30 days post-randomization)
Oral Assessment Score | Oral assessment scores will be assessed daily from the date of randomization until discharge from the ICU (up to 30 days post-randomization)
Duration of ICU and hospital stay | Subjects will be followed for these outcomes for the duration of their hospital stay up to 4 weeks after discharge from the ICU
ICU and hospital mortality | Subjects will be followed for these outcomes for the duration of their hospital stay up to 4 weeks after discharge from the ICU
Antimicrobial utilization | Utilization of antimicrobials will be assessed daily from the date of randomization until discharge from the ICU (up to 30 days post-randomization)
Acquisition of antimicrobial resistant organisms | Subjects will be followed for this outcome from the date of randomization until discharge from the ICU (up to 30 days post-randomization)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zuege, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Health Services, Calgary, Alberta, Canada